CLINICAL TRIAL: NCT00317694
Title: A Multicentre Phase II Study With Magnesium Iron Hydroxycarbonate: an Open-label, Dose-ranging Phase Followed by a Placebo-controlled, Double-blind, Parallel-group Comparison in Haemodialysis Subjects With Hyperphosphataemia
Brief Title: Efficacy and Safety Study of Magnesium Iron Hydroxycarbonate for the Reduction of High Blood Phosphate in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ineos Healthcare Limited (Industry)
Responsible Party: Chief Medical Officer, Ineos Healthcare Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IH 001 (ACT 2)
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Kidney Failure
Keywords: Hyperphosphatemia; Phosphate binder
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia | interventions — iron-magnesium hydroxycarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fermagate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fermagate — Film coated tablet 500mg
  Other Names: Magnesium iron hydroxycarbonate
  Arms: 1
Drug: Placebo — Oral administration, film coated tablet, 0mg
  Arms: 2

SUMMARY:
Magnesium iron hydroxycarbonate is a phosphate binder that absorbs phosphate from food, reducing the amount that the body can absorb.

The purpose of this study it to look at how effective and safe Magnesium iron hydroxycarbonate is in controlling levels of phosphate in the blood in patients who receive hemodialysis.

DETAILED DESCRIPTION:
High levels of phosphate in the blood are linked with serious effects, due to calcium imbalances (high levels of parathyroid hormone (PTH), bone disease, formation of calcium deposits in the body, and blood-vessel disease).

Current guidelines indicate that blood phosphorus levels should be maintained between 1.13 to 1.78 mmol/L in patients who receive hemodialysis.

This study is designed to investigate magnesium iron hydroxycarbonate's ability to lower and control patients' blood phosphate to the recommended levels and compare the average blood phosphate, calcium, calcium-phosphate product, PTH and magnesium concentrations and overall safety with placebo (or "dummy") tablets.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects on active haemodialysis, aged 18 years or over.
* Written informed consent given.
* On a stable haemodialysis regimen (three times per week) for at least 3 months and be unlikely to change their dialysis prescription during the study period.
* On a stable dose of a phosphate binder for at least 1 month prior to screening.
* Willing to abstain from taking any phosphate binder or oral magnesium, aluminum or iron-containing products and preparations, other than the study medication.
* Willing to avoid any intentional changes in diet such as fasting, dieting or overeating.
* Willing to maintain their usual type and dose of Vitamin D supplementation.

Exclusion Criteria:

* Participation in any other clinical trial using an investigational product or device within the previous 4 months.
* A significant history of alcohol, drug or solvent abuse in the opinion of the investigator.
* Any disease or condition, physical or psychological, which in the opinion of the investigator would compromise the safety of the subject or increase the likelihood of the subject being withdrawn.
* Clinically significant laboratory findings (for this subject population) in the opinion of the investigator.
* Any malignancy requiring treatment within 5 years of screening with the exception of basal cell carcinoma and Bowen's disease.
* A history of a motility disorder of the intestines, including, but not limited to, gastroparesis, ileus, pseudo-obstruction, megacolon, or mechanical obstruction.
* A significant illness in the 4 weeks before screening.
* Taking medication prescribed for seizures.
* A history of haemochromatosis.
* A history of high serum ferritin concentration of ≥ 1000ng/ml (excluding transient, treatment-induced ferritin elevation).
* A history of dysphagia or swallowing disorders that might limit the subject's ability to swallow study medication in the opinion of the investigator.
* Female subjects who are lactating or pregnant. Women of childbearing potential (pre-menopausal and not surgically sterilized) unless they are using a reliable contraceptive method, that is, barrier methods, hormones or intrauterine device.
* Current haemoglobin concentration of < 10.00 g/dL.
* Allergy to the IMP or its constituents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve controlled serum phosphate concentrations during the double-blind comparative phase | Mean of last two serum phosphate values in the double blind phase

SECONDARY OUTCOMES:
Change from baseline in mean serum phosphate concentration | Mean of last two serum phosphate values
Change from baseline in serum calcium | Specified visits throughout the study period
Change from baseline calcium-phosphate product | Specified visits throughout the study period
Change from baseline PTH | Specified visits throughout the study period
Change from baseline magnesium | Specified visits throughout the study period
Assessment of adverse events | Throughout the study period
Assessment of routine safety laboratory parameters | Specified visits throughout the study period
Assessment of physical examination | At screen and follow-up
Assessment of 12-lead electrocardiogram | At screen and follow-up
Assessment of bowel habits | Specified visits throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Simon Roe, MB ChB, Principal Investigator — Nottingham Renal and Transplant Unit, Nottingham City Hospital
Locations (15):
- United States (4):
  - 1614 West 42nd Street, Pine Bluff, Arkansas
  - US Renal Care, Stuttgart, Arkansas
  - Davita Dialysis Center, Charlotte, North Carolina
  - Southeast Renal Associates, Charlotte, North Carolina
- United Kingdom (11):
  - Renal Unit, Birmingham Heartlands Hospital, Birmingham
  - St Lukes Hospital, Bradford
  - Richard Bright Renal Unit, Southmead Hospital, Bristol
  - Addenbrookes Dialysis Centre, Addenbrookes Hospital, Cambridge
  - Renal Unit, Leicester General Hospital, Leicester
  - Dialysis Unit, Broad Green Hospital, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - General Medicine and Nephrology, Norfolk and Norwich University Hospital, Norwich
  - Nottingham Renal and Transplant Unit, Nottingham City Hospital, Nottingham
  - Sheffield Kidney Unit, Northern General Hospital, Sheffield
  - Dept. of Nephrology, Morriston Hospital, Swansea

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086